CLINICAL TRIAL: NCT01022632
Title: A Randomized, Active Controlled, Open Label, Parallel Group Study to Compare the Efficacy of Extract of Curcuma Longa (Turmeric) With Fluoxetine and to Study Its Effect as an Add on Therapy to Fluoxetine in Patients of Depression
Brief Title: Effect of Curcumin as Nutraceutical in Patients of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Bhavnagar (Other)
Collaborators: Health and Family Welfare Department, Government of Gujarat, India (Unknown); Arjuna Natural Extracts Ltd. (Industry)
Responsible Party: Dr. C. B. Tripathi, Professor and Head , Department of Pharmacology, Government Medical College, Bhavnagar-364001, Gujarat, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pharmacol no.01 /2008 Research
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Curcumin; Fluoxetine

ARMS (3):
- Fluoxetine (Active Comparator): Fluoxetine : 20 mg Once a day in morning after taking food for 6 weeks
  Interventions: Drug: Fluoxetine
- Curcumin (Experimental): Curcumin 500 mg 12 hourly after taking food in morning and evening for 6 weeks
  Interventions: Dietary Supplement: Curcumin
- Curcumin and Fluoxetine (Experimental): Curcumin 500 12 hourly after taking food in morning and evening and Fluoxetine 20 mg Once a day in morning after taking food for 6 weeks
  Interventions: Dietary Supplement: Curcumin and Fluoxetine

INTERVENTIONS:
Dietary Supplement: Curcumin — Curcumin 500 mg 12 hourly after taking food in morning and evening for 6 weeks
  Arms: Curcumin
Drug: Fluoxetine — Fluoxetine ; 20 mg Once a day in morning after taking food for 6 weeks
  Arms: Fluoxetine
Dietary Supplement: Curcumin and Fluoxetine — Curcumin 500 12 hourly after taking food in morning and evening and Fluoxetine 20 mg Once a day in morning after taking food for 6 weeks
  Arms: Curcumin and Fluoxetine

SUMMARY:
The purpose of this study is to find the effect of commonly used nutraceutical curcumin ( extract of Curcuma longa, commonly called 'Haldi' in Hindi) in patients of depression.

ELIGIBILITY:
Inclusion Criteria:

* Depression as diagnosed under DSM-IV Axis I Disorders.
* Score greater than 7 but less then 35 on the 17-item Hamilton Depression (HAM-D) Scale at screening.
* The patient has relative(s) to care for him/her
* Informed consent obtained from the patient or relative

Exclusion Criteria:

* Scores greater than 2 on the "suicide" item of HAM-D, or history of suicide attempt(s) in the past 12 months.
* Current suicidal or homicidal risk, as determined by the investigator.
* Clinically significant liver disease (such as hepatitis, cirrhosis, etc); or clinically significant elevation of liver enzyme tests (two times the upper limit of normal.
* History of seizure disorder (other than febrile).
* Patient who has had monoamine oxidase inhibitor , any selective serotonin reuptake inhibitor or any other antidepressant in last 15 days
* Any of the following DSM-IV diagnoses current (within past 3 months) schizophrenia, schizo-affective, or other psychotic disorder; bipolar disorder; current panic disorder or obsessive compulsive disorder; history of psychotic features of affective disorder (mood congruent or incongruent)
* Patient with history of untreated or unstable thyroid disorder
* Failed to respond to at least two adequate antidepressant trials (defined as 6 weeks or more treatment with either greater than or equal to 150 mg imipramine, or tricyclic equivalent), or greater than or equal to 60 mg of phenelzine, or MAOI equivalent, or greater than or equal to 100 mg of sertraline, or its SSRI equivalent.
* Have had other investigational drugs within 30 days or other psychotropic medication within 21 days.
* Known allergy or hypersensitivity to the study medications.
* Receiving psychotherapies which are specifically designed to treat depression, eg, interpersonal psychotherapy during the study period.
* Mental retardation or cognitive impairment, or any disorder that might interfere with their ability to give consent or follow study procedures and requirements.
* In case of female patients, Abstinence or effective method of contraception throughout the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Response rate according to HAM-D17 scale | 6 weeks
Mean change in HAM-D17 score | Six weeks

SECONDARY OUTCOMES:
Clinical global impression assessment | Six Weeks
Global efficacy at the end of study | Six weeks
Change in laboratory parameters (routine hematology and urine) | Six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Bharat Panchal, MD, Principal Investigator — Professor and Head, Department of Psychiatry, Sir T. General Hospital and Government Medical College, Bhavnagar-364001, Gujarat, India
Locations (1):
- Sir Takthasinhji General Hospital, Bhavnagar, Gujarat, India